CLINICAL TRIAL: NCT02225470
Title: An Open-label Randomized Parallel Two-arm Multicenter Study of Eribulin Versus Vinorelbine in Female Subjects With Locally Recurrent or Metastatic Breast Cancer, Previously Treated With At Least Two and a Maximum of Five Prior Chemotherapy Regimens, Including an Anthracycline and a Taxane
Brief Title: Eribulin Versus Vinorelbine in Subjects With Locally Recurrent or Metastatic Breast Cancer Previously Treated With Anthracyclines and Taxanes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-C086-304
Record Dates: First submitted 2014-08-05; First posted 2014-08-26 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2017-12

CONDITIONS: HER2-Negative Breast Cancer; Triple Negative Breast Cancer; Breast Cancer; Cancer of Breast; Breast Tumors
Keywords: Locally Recurrent or Metastatic Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — eribulin; Vinorelbine

ARMS (2):
- Arm A, E7389 (Eribulin Mesylate) (Experimental): The eribulin mesylate dose will be 1.4 mg/m2 administered as an intravenous bolus over 2 to 5 minutes on Days 1 and 8 of each 21-day cycle.
  Interventions: Drug: E7389 (Eribulin Mesylate)
- Arm B, Vinorelbine injection (Active Comparator): The vinorelbine dose will be 25 mg/m2 administered as an intravenous bolus on Days 1, 8, and 15 of each 21-day treatment cycle.
  Interventions: Drug: Vinorelbine injection

INTERVENTIONS:
Drug: E7389 (Eribulin Mesylate)
  Arms: Arm A, E7389 (Eribulin Mesylate)
Drug: Vinorelbine injection
  Arms: Arm B, Vinorelbine injection

SUMMARY:
This study is designed as an open-label randomized parallel two-arm multicenter efficacy, pharmacokinetics and safety study of intravenously administered eribulin versus intravenously administered vinorelbine in Chinese population. Eligible female subjects will have measurable disease according to RECIST 1.1 with the modification that chest x-ray cannot be used for assessment of disease.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study.

1. Female subjects with histologically or cytologically confirmed carcinoma of the breast:
2. Subjects with locally recurrent or metastatic disease who have received at least two, and a maximum of five, prior chemotherapeutic regimens for breast cancer, at least two of which were administered for treatment of locally recurrent or metastatic disease. Prior therapy must be documented by the following criteria prior to entry onto study:

   1. Regimens must have included an anthracycline (e.g., doxorubicin, epirubicin), and a taxane (e.g., paclitaxel, docetaxel) in any combination or order. Prior treatment with any of these agents is not required if the agents are contraindicated for a prospective subject and documented in her medical history.
   2. Some of these regimens may have been administered as adjuvant and/or neoadjuvant therapy, but at least two must have been given for locally recurrent or metastatic disease.
   3. Subjects must have proven refractory to the most recent chemotherapy as documented by progression on or within 6 months of their last chemotherapy.
   4. Subjects with Her2/neu positive tumors may also have been treated with any Her2/neu targeted agents including antibodies, small compounds or investigational drugs.
   5. Subjects may also have been treated with antihormonal therapy.
3. Have measurable disease meeting the following criteria:

   1. At least one lesion of greater than or equal to 1.0 cm in the longest diameter for a non-lymph node, or greater than or equal to 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI). If there is only one target lesion and it is a non-lymph node, it should have a longest diameter of greater than or equal to 1.5 cm.
   2. Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease based upon RECIST 1.1 to be used as a target lesion.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
5. Life expectancy of greater than or equal to 3 months.
6. subjects greater than or equal to 18 years old Age and less than or equal to 70 years old at the time of informed consent.
7. Adequate renal function as evidenced by serum creatinine less than or equal to 2.0 mg/dL or calculated creatinine clearance greater than or equal to 40 mL/min per the Cockcroft and Gault formula.
8. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L, hemoglobin greater than or equal to 10.0 g/dL, and platelet count greater than or equal to 100 x 10^9/L.
9. Adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limits of normal (ULN); and alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3.0 times ULN (in the case of liver metastases less than or equal to 5.0 times ULN).
10. Subject willing and able to comply with the study protocol for the duration of the study.
11. All female subjects will be considered to be of child-bearing potential unless they are postmenopausal (at least 12 months consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically (i.e., bilateral tubal ligation greater than or equal to 1 menstrual cycle prior to randomization, or have undergone a hysterectomy and/or bilateral oophorectomy).

    Female subjects of child-bearing potential must agree to use two forms of highly effective contraception from the last menstrual period prior to randomization (or use a double barrier method as described below until they are on two forms of highly effective contraception for at least one menstrual cycle), during study treatment, and for 3 months after the final dose of study treatment. Female subjects exempt from this requirement are subjects who practice total abstinence. If currently abstinent, the subject must agree to use a double barrier method of contraception, i.e. condom and occlusive cap (diaphragm or cervical/vault caps) with spermicide or until they are on two forms of highly effective contraception for at least one menstrual cycle if they become sexually active during study treatment and for 3 months after the final dose of study treatment. Highly effective contraception includes:
    1. Placement of intrauterine device or system,
    2. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) with spermicide,
    3. Established hormonal contraceptive methods: oral, injectable or implant. Female subjects who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product from the last menstrual period prior to randomization, and must continue to use the same hormonal contraceptive product during study treatment, and for 3 months after the final dose of study treatment,
    4. Vasectomized partner with confirmed azoospermia.
12. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol, with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Subjects who have received any of the following treatments within the specified period before treatment start:

   1. Vinorelbine has been administrated as neoadjuvant or adjuvant therapy within one year.
   2. Chemotherapy, radiation, Her2/neu targeted agents including trastuzumab or hormonal therapy within three weeks.
   3. Any investigational drug within four weeks.
   4. Blood transfusion, blood preparations and hematopoietic factor preparations such as G-CSF within two weeks.
2. Subjects of advanced breast cancer with vinorelbine effective therapy to CR/PR/SD, and PD occurred after vinorelbine discontinuing within 6 months.
3. Subjects with ineffective prior vinorelbine treatment.
4. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
5. Subjects with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least four weeks before starting treatment in this study. Any signs (e.g., radiologic) and/or symptoms of brain metastases must be stable for at least four weeks before starting study treatment; and radiographic stability should be determined by comparing a contrast-enhanced CT or MRI brain scan performed during screening to a prior scan performed at least four weeks earlier.
6. Subjects with meningeal carcinomatosis.
7. Woman must not be pregnant as documented by a negative beta-human chorionic gonadotropin (beta-hCG) test with a minimum sensitivity 25 IU/L, or equivalent unit of beta-hCG, at Screening and Baseline; nor breastfeeding.
8. Severe/uncontrolled intercurrent illness/infection.
9. Significant cardiovascular impairment (history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia).
10. Subjects with organ allografts requiring immunosuppression therapy.
11. Subjects with known positive HIV status.
12. Subjects who have had a prior malignancy, other than breast cancer, carcinoma in situ of the cervix, or non-melanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated at least five years previously with no subsequent evidence of recurrence.
13. Subjects with preexisting neuropathy greater than Grade 2.
14. Subjects with a hypersensitivity to halichondrin B and/or a halichondrin B chemical derivative.
15. Subjects who participated in a prior eribulin clinical trial whether or not eribulin was received.
16. Known intolerance to eribulin or vinorelbine (or any of the excipients).
17. Any medical condition that in the investigator's opinion may preclude subject from being entered in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) of Eribulin Arm by tumor assessment : Time to disease progression | Baseline until date of recorded disease progression or death, or up to 2 years
Progression-Free Survival (PFS) of Vinorelbine Arm by tumor assessment: Time to disease progression | Baseline until date of recorded disease progression or death, or up to 2 years
Maximum observed plasma concentration (Cmax) of Eribulin Arm in a minimum of 15 subjects | Day 1 and Day 8
Time at which the highest drug concentration occurs (tmax) of Eribulin Arm in a minimum of 15 subjects | Day 1 and Day 8
Area under the plasma concentration-time curve (AUC) of Eribulin Arm in a minimum of 15 subjects | Day 1 and Day 8
Terminal phase rate constant (lambda Z) of Eribulin Arm in a minimum of 15 subjects | Day 1 and Day 8
Terminal elimination phase half-life (t1/2) of Eribulin Arm in a minimum of 15 subjects | Day 1 and Day 8
Distribution volume at steady-state (Vss) of Eribulin Arm in a minimum of 15 subjects | Day 1 and Day 8
Total clearance (CL) of Eribulin Arm in a minimum of 15 subjects | Day 1 and Day 8

SECONDARY OUTCOMES:
Overall Survival (OS) | Baseline until date of death, or up 5 years
Duration of Response | Baseline until date of recorded disease progression or death or up to 5 years
Objective Response Rate (ORR) | Baseline until date of recorded disease progression or death, or up to 5 years
Evaluate safety parameters such as electrocardiograms | Baseline until date of recorded disease progression or death
Evaluate safety assessments parameters such as vital signs( VS) | Baseline until date of recorded disease progression or death
Evaluate safety parameters such as adverse events (AEs) | Baseline until date of recorded disease progression or death
Evaluate safety parameters such as laboratory measurements | Baseline until date of recorded disease progression or death

CONTACTS AND LOCATIONS:
Locations (35):
- China (35):
  - 04 Eisai Trial Site, Bengbu, Anhui
  - 37 Eisai Trial Site, Hefei, Anhui
  - 01 Eisai Trial Site, Beijing, Beijing Municipality
  - 03 Eisai Trial Site, Beijing, Beijing Municipality
  - 33 Eisai Trial Site, Beijing, Beijing Municipality
  - 35 Eisai Trial Site, Beijing, Beijing Municipality
  - 07 Eisai Trial Site, Fuzhou, Fujian
  - 08 Eisai Trial Site, Fuzhou, Fujian
  - 20 Eisai Trial Site, Guangzhou, Guangdong
  - 36 Eisai Trial Site, Guangzhou, Guangdong
  - 10 Eisai Trial Site, Nanning, Guangxi
  - 12 Eisai Trial Site, Shijiazhuang, Hebei
  - 11 Eisai Trial Site, Harbin, Heilongjiang
  - 38 Eisai Trial Site, Zhengzhou, Henan
  - 14 Eisai Trial Site, Wuhan, Hubei
  - 15 Eisai Trial Site, Wuhan, Hubei
  - 05 Eisai Trial Site, Changsha, Hunan
  - 13 Eisai Trial Site, Changsha, Hunan
  - 34 Eisai Trial Site, Changsha, Hunan
  - 18 Eisai Trial Site, Nanjing, Jiangsu
  - 31 Eisai Trial Site, Nanjing, Jiangsu
  - 16 Eisai Trial Site, Changchun, Jilin
  - 17 Eisai Trial Site, Changchun, Jilin
  - 06 Eisai Trial Site, Dalian, Liaoning
  - 19 Eisai Trial Site, Shenyang, Liaoning
  - 21 Eisai Trial Site, Yinchuang, Ningxia
  - 24 Eisai Trial Site, Xi'an, Shaanxi
  - 28 Eisai Trial Site, Xi'an, Shaanxi
  - 22 Eisai Trial Site, Qingdao, Shandong
  - 09 Eisai Trial Site, Shanghai, Shanghai Municipality
  - 23 Eisai Trial Site, Taiyuan, Shanxi
  - 26 Eisai Trial Site, Chengtu, Sichuan
  - 27 Eisai Trial Site, Tianjin, Tianjin Municipality
  - 30 Eisai Trial Site, Yunnan, Yunnan
  - 40 Eisai Trial Site, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Yuan P, Hu X, Sun T, Li W, Zhang Q, Cui S, Cheng Y, Ouyang Q, Wang X, Chen Z, Hiraiwa M, Saito K, Funasaka S, Xu B. Eribulin mesilate versus vinorelbine in women with locally recurrent or metastatic breast cancer: A randomised clinical trial. Eur J Cancer. 2019 May;112:57-65. doi: 10.1016/j.ejca.2019.02.002. Epub 2019 Mar 29. PMID 30928806